CLINICAL TRIAL: NCT07297979
Title: A Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Xaluritamig in Adult, Adolescent and Pediatric Participants With Relapsed or Refractory Ewing Sarcoma
Brief Title: Evaluation of Xaluritamig in Adults, Adolescents and Children With Relapsed or Refractory Ewing Sarcoma (EWS)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 20200034
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ewing Sarcoma
Keywords: Relapsed or refractory Ewing sarcoma; EWS; Xaluritamig; AMG 509
MeSH Terms: conditions — Sarcoma, Ewing; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Dose Confirmation) (Experimental): Part 1 will begin with a pre-specified xaluritamig target dose and frequency. Multiple dose levels and/or alternative dose regimens may be explored in parallel to determine 1 or more recommended doses for expansion, which is/are considered safe, based on emerging data.
  Interventions: Drug: Xaluritamig
- Part 2 (Dose Expansion) (Experimental): Participants will be treated in Part 2 after the recommended doses for expansion for xaluritamig are determined in Part 1 to further characterize preliminary antitumor activity and safety.
  Interventions: Drug: Xaluritamig

INTERVENTIONS:
Drug: Xaluritamig — Participants will receive xaluritamig via short-term intravenous (IV) infusion.
  Other Names: AMG 509

SUMMARY:
The main objectives of this trial are to determine the recommended dose for expansion of xaluritamig (dose confirmation part only) and to determine the safety and tolerability of xaluritamig in adult, adolescent and pediatric participants with relapsed or refractory EWS.

ELIGIBILITY:
Inclusion Criteria:

1. Part 1: evaluable disease as defined by RECIST v1.1, as determined by the site investigator.

   Part 2: measurable disease as defined by RECIST v1.1, as determined by the site investigator.
2. Histologically or cytologically confirmed EWS with molecular evidence of an EWSR1 translocation with an E26 transformation-specific (ETS) family gene, eg, FLI1, ETS-related gene [ERG]) via next generation sequencing (based on local testing).
3. Relapsed or refractory EWS following at least 1 line of chemotherapy (including treatment with an anthracycline and at least 1 alkylating agent).
4. Performance status:

   1. Karnofsky ≥ 70% for participants ≥ 16 years of age.
   2. Lansky ≥ 70% for participants < 16 years of age.
5. Adequate organ function, defined as follows:

   a. Hematological function: i. Absolute neutrophil count ≥ 1.0 x 109/L, provided that:
   * the participant has not received short-acting growth factor support within 7 days before screening assessment, and
   * the participant has not received long-acting growth factor support within 14 days before screening assessment.

   ii. Platelet count ≥ 75 x 109/L, provided that:
   * the participant has not received a platelet transfusion within 7 days before screening assessment, and
   * the participant has not received a platelet stimulating agent within 14 days before screening assessment.

     b. Renal function: i. Estimated glomerular filtration rate based on Modification of Diet in Renal Disease (MDRD) calculation ≥ 30 mL/min/1.73 m^2 for participants ≥ 18 years of age.

   ii. estimated glomerular filtration rate based on Schwartz (2009) calculation ≥ 30 mL/min/1.73 m^2 for participants < 18 years of age.

   c. Hepatic function: i. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (or ≤ 5 x ULN for participants with liver metastases).

   ii. Total bilirubin (TBL) ≤ 1.5 x ULN (unless related to Gilbert's or Meulengracht disease).

   d. Pulmonary function: i. Baseline oxygen saturation > 92% in room air at rest and no oxygen supplementation.

   e. Cardiac function: i. Left ventricular ejection fraction ≥ 50%. If left ventricular ejection fraction cannot be measured, then left ventricular fractional shortening ≥ 28%.
6. Participants of childbearing potential must use protocol-specified contraception to prevent pregnancy during treatment and for an additional 6 months after the last dose of xaluritamig.

Exclusion Criteria:

1. Untreated central nervous system (CNS) metastases or leptomeningeal disease. Participants with a history of treated CNS metastases are eligible if there is radiographic evidence of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.
2. History of other malignancy within the past 2 years, except for malignancy treated with curative intent with low risk for recurrence (approximately < 10%) and with no known active disease present for >1 year before enrollment.
3. Active autoimmune disease that has required systemic treatment (except physiologic adrenal hormone replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study. Participants with Type 1 diabetes, vitiligo, psoriasis, hypo- or hyper-thyroid disease not requiring immunosuppressive treatment are permitted.
4. Participants who received anti-cancer therapy administered within the following minimum washout periods prior to first dose of xaluritamig:

   1. Cytotoxic chemotherapy: 21 days.
   2. Small molecules including tyrosine kinase inhibitors: 7 days or 5 half-lives, whichever is shorter.
   3. Monoclonal antibodies, immune checkpoint inhibitors, bispecific antibodies and other biologic agents: 28 days or 5 half-lives, whichever is shorter.
   4. Cellular therapies including Chimeric Antigen Receptor T-cell therapy (CAR-T), adoptive T-cell therapy: 56 days.
   5. Radiotherapy: 14 days for focal therapy, 28 days for large field therapy or involving > 30% of the bone marrow.
   6. Stem cell transplant: 12 weeks for autologous, 6 months for allogeneic, with no active graft-versus-host disease.
   7. Any other therapy or investigational agent: 28 days or 5 half-lives, whichever is longer.
5. Requirement for chronic systemic corticosteroid therapy (prednisone dose > 10 mg/day [> 0.25 mg/kg/day if < 40 kg] or equivalent) or any other immunosuppressive therapies (including anti-tumour necrosis factor α (TNFα) therapies) unless stopped (with adequate tapering) within 28 days before first dose of xaluritamig.
6. Currently pregnant (confirmed with positive pregnancy test) or breastfeeding or planning to become pregnant, donate eggs, or breastfeed while on trial until an additional 6 months after the last dose of trial intervention.
7. Unwilling to abstain from donating sperm during treatment and for an additional 6 months after the last dose of xaluritamig.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-22 (Estimated); Primary Completion 2030-04-29 (Estimated); Study Completion 2030-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing a Dose-limiting Toxicity (DLT) (Part 1 Only) | Up to 42 days
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 2.5 years
  This includes treatment-emergent, treatment-related, serious, and fatal adverse events. Any changes in safety assessments (vital signs and clinical laboratory tests) will be recorded as adverse events.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of Xaluritamig | Up to approximately 6 months
Time to Cmax (tmax) of Xaluritamig | Up to approximately 6 months
Minimum Serum Concentration (Cmin) of Xaluritamig | Up to approximately 6 months
Accumulation Following Multiple Doses of Xaluritamig | Up to approximately 6 months
Serum Concentration Before Dosing (Ctrough) of Xaluritamig | Up to approximately 6 months
Half-life (t½) of Xaluritamig | Up to approximately 6 months
Area Under the Serum Concentration-time Curve (AUC) of Xaluritamig | Up to approximately 6 months
Confirmed Objective Response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 6 months
Disease Control per RECIST v1.1 | Up to approximately 6 months
Time to Response (TTR) per RECIST v1.1 | Up to approximately 6 months
Duration of Confirmed Response (DOR) per RECIST v1.1 | Up to approximately 6 months
Progression-free Survival (PFS) per RECIST v1.1 | Up to approximately 6 months
Time to Progression (TTP) per RECIST v1.1 | Up to approximately 6 months
Time to First Subsequent Anti-cancer Therapy | Up to approximately 6 months
Overall Survival (OS) | Up to approximately 2 years
Number of Participants with Anti-xaluritamig Antibody Formation | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com